CLINICAL TRIAL: NCT05516264
Title: Behavioural and Physiological Responses to Dog Visits in Nursing Homes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ANIMAL CONTACT 4
Record Dates: First submitted 2022-08-19; First posted 2022-08-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Physiological Responses; Behavior; Mood
Keywords: Human-animal contact; Non-invasive measure
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Participants from 2 nursing homes (25+25) are all receive three visit with a dog and three without a dog. It is randomised whter participents receive the dog visits first or last.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dog visits first (Other): Participants receive the three dogs visits first and then, after a break, receive the three control visits
  Interventions: Behavioral: Dog visits/control visits
- Control visits first (Other): Participants receive the three control visits first and then, after a break, receive the three dog visits
  Interventions: Behavioral: Control visits/dog visits

INTERVENTIONS:
Behavioral: Dog visits/control visits — See arm description above
  Arms: Dog visits first
Behavioral: Control visits/dog visits — See arm description above
  Arms: Control visits first

SUMMARY:
In brief the study aims to investigate how nursing home residents receiving dog visits respond to contact with the dog, by comparing visits with and without a dog present. The investigators will measure the response with non-invasive measures of the immediate physiological response, and objective behavioural measurements to quantity the activity and the actual amount and intensity of contact to the dog.

DETAILED DESCRIPTION:
The residents will receive six 10-minute visits, three visits with a dog and three without a dog, with a week-long break in between the two visit types. The participants will be randomly assigned to receive either the three dog visits or the three visits without a dog first. The visits will be from the same person, and the dog visits will be accompanied with the same dog each time. During dog visits, the dog will be available for touch, and the resident will be encouraged to interact with the dog.

Before each visit the resident is fitted with the equipment for measuring continuously recorded physiological measures and then relaxes for 30 minutes. Immediately before and five and 30 minutes after each visit, the investigators obtain a saliva sample to detect cortisol levels.

The behaviour of the participants will be video recorded during the visits to quantify the frequency and duration of predefined behavioural elements, using ethological methodology. The investigators will quantify the participants' activity during the visits as well as the frequency and duration of tactile contact with the dog, and verbal communication with the dog and the visitor.

In addition, the visitor and the observer present during the visit will subjectively assess the resident's perception of the visit.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 years or more
* Able to sit during visits (either in a chair or in a bed)

Exclusion Criteria:

* Known allergy to dogs
* Known fear of dogs

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart rate | During visit no. 1, from 30 minutes before the visit to 30 minutes after
  The test person wears a device placed on the upper arm
Heart rate | During visit no. 2, from 30 minutes before the visit to 30 minutes after
  The test person wears a device placed on the upper arm
Heart rate | During visit no. 3, from 30 minutes before the visit to 30 minutes after
  The test person wears a device placed on the upper arm
Heart rate | During visit no. 4, from 30 minutes before the visit to 30 minutes after
  The test person wears a device placed on the upper arm
Heart rate | During visit no. 5, from 30 minutes before the visit to 30 minutes after
  The test person wears a device placed on the upper arm
Heart rate | During visit no. 6, from 30 minutes before the visit to 30 minutes after
  The test person wears a device placed on the upper arm
Heart rate variability | During visit no. 1, from 30 minutes before the visit to 30 minutes after
  Heart rate variability is calculated from heart rate data
Heart rate variability | During visit no. 2, from 30 minutes before the visit to 30 minutes after
  Heart rate variability is calculated from heart rate data
Heart rate variability | During visit no. 3, from 30 minutes before the visit to 30 minutes after
  Heart rate variability is calculated from heart rate data
Heart rate variability | During visit no. 4, from 30 minutes before the visit to 30 minutes after
  Heart rate variability is calculated from heart rate data
Heart rate variability | During visit no. 5, from 30 minutes before the visit to 30 minutes after
  Heart rate variability is calculated from heart rate data
Heart rate variability | During visit no. 6, from 30 minutes before the visit to 30 minutes after
  Heart rate variability is calculated from heart rate data
Behaviour during visits | During visit no. 1, from 30 minutes before the visit to 30 minutes after
  The test persons behaviour is observed
Behaviour during visits | During visit no. 2, from 30 minutes before the visit to 30 minutes after
  The test persons behaviour is observed
Behaviour during visits | During visit no. 3, from 30 minutes before the visit to 30 minutes after
  The test persons behaviour is observed
Behaviour during visits | During visit no. 4, from 30 minutes before the visit to 30 minutes after
  The test persons behaviour is observed
Behaviour during visits | During visit no. 5, from 30 minutes before the visit to 30 minutes after
  The test persons behaviour is observed
Behaviour during visits | During visit no. 6, from 30 minutes before the visit to 30 minutes after
  The test persons behaviour is observed
Salivary cortisol | Visit 1, 2 minutes before visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 2, 2 minutes before visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 3, 2 minutes before visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 4, 2 minutes before visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 5, 2 minutes before visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 6, 2 minutes before visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 1, 5 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 2, 5 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 3, 5 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 4, 5 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 5, 5 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 6, 5 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 1, 30 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 2, 30 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 3, 30 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 4, 30 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 5, 30 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute
Salivary cortisol | Visit 6, 30 minutes after visit
  Saliva is obtained from the testperson with a swab which held his/her mouth for one minute

SECONDARY OUTCOMES:
The visitor's and observer's perception of how the visit was experienced by the test person. | 5 minutes after visit 1
  Minimum value 0 (worst possible visit) to 100 (best possible visit)
The visitor's and observer's perception of how the visit was experienced by the test person. | 5 minutes after visit 2
  Minimum value 0 (worst possible visit) to 100 (best possible visit)
The visitor's and observer's perception of how the visit was experienced by the test person. | 5 minutes after visit 3
  Minimum value 0 (worst possible visit) to 100 (best possible visit)
The visitor's and observer's perception of how the visit was experienced by the test person. | 5 minutes after visit 4
  Minimum value 0 (worst possible visit) to 100 (best possible visit)
The visitor's and observer's perception of how the visit was experienced by the test person. | 5 minutes after visit 5
  Minimum value 0 (worst possible visit) to 100 (best possible visit)
The visitor's and observer's perception of how the visit was experienced by the test person. | 5 minutes after visit 6
  Minimum value 0 (worst possible visit) to 100 (best possible visit)
Visual analoque scale of the testpersons' evaluation of the visit | 5 minutes after visit 1
  Minimum value 0 (worst possible experience) to 100 (best possible experience)
Visual analoque scale of the testpersons' evaluation of the visit | 5 minutes after visit 2
  Minimum value 0 (worst possible experience) to 100 (best possible experience)
Visual analoque scale of the testpersons' evaluation of the visit | 5 minutes after visit 3
  Minimum value 0 (worst possible experience) to 100 (best possible experience)
Visual analoque scale of the testpersons' evaluation of the visit | 5 minutes after visit 4
  Minimum value 0 (worst possible experience) to 100 (best possible experience)
Visual analoque scale of the testpersons' evaluation of the visit | 5 minutes after visit 5
  Minimum value 0 (worst possible experience) to 100 (best possible experience)
Visual analoque scale of the testpersons' evaluation of the visit | 5 minutes after visit 6
  Minimum value 0 (worst possible experience) to 100 (best possible experience)

CONTACTS AND LOCATIONS:
Locations (1):
- Karen Thodberg, Højslev, Denmark

IPD SHARING:
Plan to Share IPD: No